CLINICAL TRIAL: NCT03228017
Title: Subclinical Cardiovascular Disease in Psoriatic Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 17-00692
Record Dates: First submitted 2017-07-11; First posted 2017-07-24 (Actual); Results first posted 2021-09-28 (Actual); Last update posted 2021-09-28 (Actual); Status verified 2021-08

CONDITIONS: Cardiovascular Diseases; Myocardial Infarction; Atherosclerotic Cardiovascular Disease; Thrombotic Vascular Disease
Keywords: cardiovascular disease; CVD
MeSH Terms: conditions — Cardiovascular Diseases; Myocardial Infarction; Atherosclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Psoriatic Disease Patients (Other): Moderate to severe psoriatic disease
  Interventions: Drug: Aspirin and/or Atorvastatin
- Healthy Control (No Intervention)

INTERVENTIONS:
Drug: Aspirin and/or Atorvastatin — This follow-up will allow us to assess how aspirin and/or atorvastatin affect platelet and endothelial function and inflammation.
  Arms: Psoriatic Disease Patients

SUMMARY:
This study will look at how chronic inflammation seen in psoriatic disease translates into the increased atherosclerotic and thrombotic risk and how treatment reduces this CVD risk. The Aim of this study is to 1) Evaluate the association between moderate to severe psoriatic disease and measures of vascular function. 2) Evaluate the association between moderate to severe psoriatic disease and measures of thrombotic risk. 3) Understand how traditional medications used in cardiovascular disease (CVD) prevention such as aspirin and statins affect vascular function and thrombotic risk in those with moderate to severe psoriatic disease.

DETAILED DESCRIPTION:
Cardiovascular disease (CVD) remains the leading cause of death in the US. Five modifiable risk factors: smoking, hyperlipidemia, diabetes, hypertension and obesity, account for 50% of CVD mortality between the ages of 45 - 79.1 These traditional cardiac risk factors dictate who to treat with primary prevention measures but do not take into account patient-specific disease states such as psoriatic disease including psoriasis and psoriatic arthritis, which predispose to chronic inflammation. Patients with psoriatic disease have an increased risk of atherosclerotic heart disease and myocardial infarctions compared to matched controls.

ELIGIBILITY:
Inclusion Criteria:

* Subjects with a history of moderate to severe psoriatic disease
* Group 2: Healthy subjects without known psoriatic disease or cardiovascular disease

Exclusion Criteria:

* Unable to speak Spanish or English
* Active smoking (within the past year)
* Autoimmune, rheumatologic or inflammatory disease which are not psoriasis or psoriatic arthritis
* Known active cancer receiving treatment
* Pregnancy
* Anemia (hemoglobin < 9 mg/dl) or thrombocytopenia (Platelet count <75), or thrombocytosis (Platelet count >600)
* A history of severe bleeding or bleeding disorders
* Current medication use which interact with either aspirin or atorvastatin
* Chronic kidney disease (CrCl < 30ml/min)
* Congestive heart failure
* Currently taking aspirin or a statin.
* NSAID use within the past 48 hours

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2017-08-01 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2019-04-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Berger, MD, Principal Investigator — NYU Langone Health
Locations (1):
- New York University School of Medicine, New York, New York, United States

REFERENCES:
- [Derived] Garshick MS, Block R, Drenkova K, Tawil M, James G, Brenna JT. Statin therapy upregulates arachidonic acid status via enhanced endogenous synthesis in patients with plaque psoriasis. Prostaglandins Leukot Essent Fatty Acids. 2022 May;180:102428. doi: 10.1016/j.plefa.2022.102428. Epub 2022 Apr 16. PMID 35490599
- [Derived] Garshick MS, Tawil M, Barrett TJ, Salud-Gnilo CM, Eppler M, Lee A, Scher JU, Neimann AL, Jelic S, Mehta NN, Fisher EA, Krueger JG, Berger JS. Activated Platelets Induce Endothelial Cell Inflammatory Response in Psoriasis via COX-1. Arterioscler Thromb Vasc Biol. 2020 May;40(5):1340-1351. doi: 10.1161/ATVBAHA.119.314008. Epub 2020 Mar 5. PMID 32131611
- [Derived] Garshick MS, Barrett TJ, Wechter T, Azarchi S, Scher JU, Neimann A, Katz S, Fuentes-Duculan J, Cannizzaro MV, Jelic S, Fisher EA, Krueger JG, Berger JS. Inflammasome Signaling and Impaired Vascular Health in Psoriasis. Arterioscler Thromb Vasc Biol. 2019 Apr;39(4):787-798. doi: 10.1161/ATVBAHA.118.312246. PMID 30760013

RESULTS

PARTICIPANT FLOW:
Groups:
- Healthy Control: Healthy Control
Period: Overall Study
Arm/Group | Psoriatic Disease Patients | Healthy Control
Started | 45 | 18
Completed | 45 | 18
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Psoriatic Disease Patients | Healthy Control | Total
Number analyzed (Participants) | 45 | 18 | 63
Age, Continuous [Mean (Standard Deviation); unit: years] | 45 (14.2) | 40.5 (12.7) | 42.75 (13.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 8 | 31
  Male | 22 | 10 | 32
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4 | 2 | 6
  Not Hispanic or Latino | 38 | 15 | 53
  Unknown or Not Reported | 3 | 1 | 4
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 3 | 2 | 5
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 2 | 3 | 5
  White | 37 | 12 | 49
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 3 | 1 | 4
Region of Enrollment [Number; unit: participants]
  United States | 45 | 18 | 63

OUTCOME MEASURES:

1. Primary Outcome: Mean Fold Change in Brachial Vein Endothelial Inflammatory Transcript
Description: Endothelial sampling coupled to real-time PCR analysis will be used to monitor brachial vein endothelial inflammation
Time Frame: Baseline, 5 Months
Measure: Mean (Standard Deviation); unit: Fold Change
Arm/Group | Psoriatic Disease Patients | Healthy Control
Number analyzed (Participants) | 45 | 18
Fold Change | 8.6 (8.6) | 2.8 (2.2)

2. Secondary Outcome: Fold Change Change in Composite Endothelial Inflammation
Description: Endothelial inflammation will be monitored after 2 weeks of aspirin 81mg therapy
Time Frame: Baseline (pre-Aspirin), 2 weeks (post-Aspirin)
Measure: Mean (Full Range); unit: Fold Change
Arm/Group | Psoriatic Disease Patients | Healthy Control
Number analyzed (Participants) | 15 | 15
Fold Change | -0.28 [-0.4 to -.15] | -0.04 [-0.17 to 0.09]

3. Secondary Outcome: Fold Change in Composite Endothelial Inflammation
Description: Endothelial inflammation will be monitored after 2- weeks of 40mg of atorvastatin therapy.
Time Frame: Baseline (pre-Atorvastatin), 2 weeks (post-Atorvastatin)
Measure: Mean (Full Range); unit: Fold Change
Arm/Group | Psoriatic Disease Patients | Healthy Control
Number analyzed (Participants) | 20 | 10
Fold Change | -0.1 [-.21 to -0.003] | 0.1 [-.04 to 0.25]

4. Secondary Outcome: Change in Levels of Circulating Thromboxane B2
Description: Platelet activation is measured by levels of circulating thromboxane b2, which will be measured after 2- weeks of aspirin 81mg therapy
Time Frame: Baseline (pre-Aspirin), 2 weeks (post-Aspirin)
Measure: Median (Standard Deviation); unit: ng/ml
Arm/Group | Psoriatic Disease Patients | Healthy Control
Number analyzed (Participants) | 15 | 15
ng/ml | 1 (0.8) | 4.05 (3)

ADVERSE EVENTS:
Time Frame: 2 weeks
Arm/Group | Psoriatic Disease Patients | Healthy Control
All-Cause Mortality (participants affected / at risk) | 0/45 | 0/18
Serious Adverse Events (participants affected / at risk) | 0/45 | 0/18
Other Adverse Events (participants affected / at risk) | 0/45 | 0/18

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-03-22): https://cdn.clinicaltrials.gov/large-docs/17/NCT03228017/Prot_SAP_000.pdf